CLINICAL TRIAL: NCT02120651
Title: Effect of the Fibrin Monomer in the Integrity of the Graft During Tympanoplasty Compared With the Effect of the Hemostatic Sponge
Brief Title: Fibrin Monomer Compared With Hemostatic Sponge in the Integrity of the Graft During Tympanoplasty
Acronym: TISSUCOL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CLOTILDE FUENTES OROZCO (Other Government)
Responsible Party: Sponsor-Investigator, CLOTILDE FUENTES OROZCO, PhD, Instituto Mexicano del Seguro Social
Organization: Instituto Mexicano del Seguro Social (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TISSUCOL-012
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Tympanic Membrane Perforation
Keywords: Fibrin monomer; Tympanoplasty; Hemostatic sponge
MeSH Terms: conditions — Tympanic Membrane Perforation | interventions — fibrinmonomer; Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fibrin monomer (Active Comparator): 40 patients, the material was ready to use in the case of the fibrin monomer it was maintained in cooling according to the indications of lab maintenance and it was taken out a few minutes before using the material to prepare it according to instructional use and thus ensure that the conditions of maintenance of equipment are appropriate to the best outcome with their use.
  Interventions: Procedure: Fibrin monomer
- Hemostatic sponge (Placebo Comparator): 40 patients, the material was ready to use in the case of the hemostatic sponge was cut into small size, prepared and impregnated with hydrocortisone as in the standard procedure.
  Interventions: Procedure: Hemostatic sponge

INTERVENTIONS:
Procedure: Fibrin monomer — Fibrin monomer by microscopic tympanoplasty, every 4 weeks up to 3 months is evaluated graft integrity by standard audiologic and tympanometric parameters.
  Other Names: Tissucol
  Arms: Fibrin monomer
Procedure: Hemostatic sponge — Hemostatic sponge by microscopic tympanoplasty, every 4 weeks up to 3 months is evaluated graft integrity by standard audiologic and tympanometric parameters.
  Arms: Hemostatic sponge

SUMMARY:
The diagnosis of tympanic perforation reaches a high number of records in otorhinolaryngology services worldwide. Most of the tympanoplasties are performed in patients whose cause of perforation and hearing loss was chronic otitis media; this entity affects the population between 0.5 to 30% , the statistics mention more than 20 million people with this disease in the world. Since the introduction of tympanoplasty in the second half of the nineteenth century there have been numerous publications nationally and internationally about various experiences and new techniques. Including the use of fibrin monomer . This procedure is usually performed with the use of hemostatic sponge and recently with fibrin monomer, both materials are part of the basic input and surgical hemostatic agents. In this hospital are performed on average 110 tympanoplasty per year which has a percentage of non- integrity of the graft in the case of microscopic tympanoplasties using hemostatic sponge of 16% which is similar to the index of lack of integrity of the graft in microscopic tympanoplasties reported worldwide (18%), with the recent addition to the service of fibrin monomer, was necessary to evaluate if this material contributes to the integrity of the graft in microscopic tympanoplasty, as it has been reported in previous studies, so if there is found more integrity with this material, it can be recommended for routine use, improving the final prognosis of the patients.

DETAILED DESCRIPTION:
Objective: Assess the effect of fibrin monomer in the integrity of the graft during tympanoplasties compared with the effect of the hemostatic sponge at the hospital of specialties Western Medical Center.

Material and Methods: Clinical trial with single blind, parallel-groups and randomized assignation. There were included patients with a diagnosis of tympanic perforation, candidates for surgical treatment by performing only microscopic tympanoplasties, which fulfilled the selection criteria. The main variable of the study was the integrity of the graft.

The statistical analysis was performed according to the nature of variables, for continuous data using measures of central tendency and dispersion and for the qualitative data with frequencies and percentages. To evaluate the effect of fibrin monomer relative to the hemostatic sponge, the data relating to the integrity of the graft between the groups were analyzed by chi-square.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with tympanic perforation and with surgical indication of Tympanoplasty (without otorrhea for 6 months)

Exclusion Criteria:

* Background of tympanic perforation caused by allergic or pulmonary diseases including asthma and allergic rhinitis.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Integrity of the graft | every 4 weeks up to 3 months
  Integrity of the graft (100%) was evaluated by standard audiologic and tympanometric parameters.

SECONDARY OUTCOMES:
Complications | every 4 weeks up to 3 months
  Adhesions, granulomas and hearing loss

CONTACTS AND LOCATIONS:
Overall Officials: Clotilde Fuentes-Orozco, PhD, Study Director — Instituto Mexicano del Seguro Social; Luis-Humberto Govea-Camacho, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Western Medical Center, Mexican Institute of Social Security, Guadalajara, Jalisco, Mexico